CLINICAL TRIAL: NCT06542289
Title: Single-Arm, Multicenter Study to Evaluate the Safety and Effectiveness of the BlinkER System in Participants With Facial Nerve Palsy
Brief Title: Safety and Effectiveness of the BlinkER System in Participants With Facial Nerve Palsy
Acronym: Paralysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurotrigger Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-CLN-00200
Record Dates: First submitted 2024-07-22; First posted 2024-08-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-11

CONDITIONS: Bell's Palsy; Ramsay Hunt Syndrome; Lyme Disease; Facial Palsy
Keywords: BlinkER System; BlinkER
MeSH Terms: conditions — Bell Palsy; Herpes Zoster Oticus; Lyme Disease; Facial Paralysis

STUDY DESIGN:
Intervention Model Description: A single-arm study for subjects diagnosed with facial nerve palsy.
Masking Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- BlinkER system treatment (Experimental): A prospective single-arm multicenter pivotal study designed to evaluate the safety and effectiveness of the BlinkER System in achieving eyelid closure in participants with facial nerve palsy. Participants will receive the NeuroTrigger Basic System and use it for up to 3 months.
  Interventions: Device: BlinkER device.

INTERVENTIONS:
Device: BlinkER device. — Participants will use the BlinkER System for 8-16 hours daily (removed during sleep) at approximately 10 blinks/minute. The stimulation cycle will be ON and OFF to achieve the desired blink rate. Participants will receive training on device usage before starting the study.

SUMMARY:
Prospective, single-arm, multicenter, single-masked, pivotal study to Evaluate the Safety and Effectiveness of the Blinker system in Participants with Facial Nerve Palsy.

DETAILED DESCRIPTION:
A single-arm, multicenter study will be conducted to evaluate the safety and effectiveness of the Blinker system in achieving eyelid closure over a 3-month period in individuals with facial nerve palsy. The study aims to enroll at least 80 participants for evaluation. Participants will use the investigative device for a duration of 3 months.

All subjects will undergo the following visits: Screening/Baseline (Day 0), Day 1, Week 1, Week 2, Month 1, Month 2 (Remote visit), and Month 3.

The inclusion criteria for participants will be unilateral facial palsy due to conditions such as Bell's palsy, Ramsay Hunt syndrome, malignant or benign tumor resection, Lyme disease, cerebrovascular accident (hemorrhagic or ischemic), or trauma.

The estimated total study duration is 12 months.

ELIGIBILITY:
Inclusion Criteria:

22 years of age or older

* Unilateral facial palsy due to any of the following: Bell's palsy, Ramsay Hunt syndrome, malignant or benign tumor resection, Lyme disease, cerebrovascular accident (hemorrhagic or ischemic), or trauma
* A deficit in eye closure during blinking, defined as a mean blink score ≤2.0 in the study eye on the scale by Mäkelä, et al, as graded by the investigator.
* Willing and able to comply with the study procedures and follow-up
* Willing and able to provide informed consent
* English, Spanish, or Hebrew, Arabic -speaking
* In a trial with the BlinkER System, the device produces blinks sufficient to cover the pupil in the study eye, defined as a mean grade ≥ 3.0 on the Mäkelä scale, as graded by the investigator.
* Participant successfully completes BlinkER System training and certification

Exclusion Criteria:

* Bilateral facial paralysis (for example Parkinson's Disease)
* History of prior intervention that is providing closure of the eyelids (e.g., facial reanimation, complete tarsorrhaphy surgery, etc.)
* Has an implanted eyelid weight in the study eyelid.
* History of diabetic neuropathy, unstable cardiovascular disease, neurologic disease causing severe cognitive or motor impairment, severe immunological deficiency, or malignant diseases that are not in remission
* Signs of corneal infection, severe ocular surface inflammation, or significant periorbital skin inflammation/infection
* Suspected or diagnosed epilepsy.
* Cancerous lesions in the area where the BlinkER system electrodes will be applied.
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device
* Cornea or iris abnormalities that preclude visualization of the pupil
* Cranial nerve V palsy or neurotrophic keratitis
* Synkinesis that results in eyelid closure
* Known allergy to any of the patient-contacting materials of the BlinkeER electrode (i.e. polyethylene (PET) film tape or hydrogel)
* Participants who are pregnant or nursing.
* Participation in another ophthalmic clinical trial within one year prior to enrollment. Participant must also be willing to refrain from another ophthalmic study for the duration of the study.
* Co-existing condition, either ocular or non-ocular that, in the judgement of the investigator could affect the safety or effectiveness of treatment or the compliance of the participant to the protocol.

Ages: 22 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The percent of participants who achieve eyelid closure graded by independent, masked graders at a reading center. | 2 weeks
  Eyelid closure is defined as a mean blink score as graded by the independent masked graders using the Mäkelä scale:
  5- Complete eye closure 4- Nearly complete eye closure 3- Eyelid covers the pupil 2-Eyelid partially covers the pupil
  1-Twitch 0- No movement

SECONDARY OUTCOMES:
Percent of participants who achieve eyelid closure in the study eye at 1 month. | up to 1 month
  Eyelid closure is defined as a mean blink score as graded by the independent masked graders using the Mäkelä scale:
  5- Complete eye closure 4- Nearly complete eye closure 3- Eyelid covers the pupil 2-Eyelid partially covers the pupil
  1-Twitch 0- No movement
Percent of participants who achieve eyelid closure in the study eye at 3 months. | up to 3 months
  Eyelid closure is defined as a mean blink score as graded by the independent masked graders using the Mäkelä scale:
  5- Complete eye closure 4- Nearly complete eye closure 3- Eyelid covers the pupil 2-Eyelid partially covers the pupil
  1-Twitch 0- No movement
safety outcome is the rate of adverse events through 3 months. | 3 months
  safety measures include IOP, BCVA, slit lamp biomicroscopy and non-mydriatic fundus findings, and VAS pain and discomfort questionnaire evaluated at the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Ben Cnaan, MD, Principal Investigator — Sourasky Medical Center - Ichilov; Alison Rand, MD, Principal Investigator — Rand Eye Institute; Jennifer Tan, MD, Principal Investigator — Sheffield Teaching Hospital - Royal Hallamshire Hospital; David Zadok, MD, Principal Investigator — Shaarei Zedek MC; Bernard Chang, MD, Principal Investigator — Leeds Teaching Hospital - St. James University Hospital; Reza Vagefi, MD, Principal Investigator — Tufts University
Locations (1):
- Rand Eye Institute, Deerfield Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No